CLINICAL TRIAL: NCT02820701
Title: Ultrasound Evaluation of the Effect of Osteopathic Manipulative Treatment on Sacral Base Asymmetry
Brief Title: Ultrasound Evaluation of OMT for Sacral Base Asymmetry
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: A.T. Still University of Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 160616-001
Record Dates: First submitted 2016-06-29; First posted 2016-07-01 (Estimated); Last update posted 2019-01-10 (Actual); Status verified 2019-01

CONDITIONS: Manipulation, Osteopathic
Keywords: Osteopathic Manipulation; Somatic Dysfunction; Musculoskeletal Ultrasound

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): All participants will receive an initial palpatory assessment of the sacral base asymmetry and then an initial ultrasound evaluation of sacral base asymmetry. After the ultrasound assessment, the control group will wait in another room for approximately 30 minutes.
- Treatment (Experimental): All participants will receive an initial palpatory assessment of the sacral base asymmetry and then an initial ultrasound evaluation of sacral base asymmetry. Participants in the Treatment group will receive OMT to address sacral base asymmetry after the initial ultrasound assessment.
  Interventions: Procedure: OMT

INTERVENTIONS:
Procedure: OMT — Osteopathic Manipulative Treatment to low back region
  Arms: Treatment

SUMMARY:
This prospective, randomized, controlled trial is proposed to investigate the effect of OMT on sacral base asymmetry as assessed by ultrasound.

DETAILED DESCRIPTION:
The proposed prospective, randomized, controlled trial will investigate the effect of osteopathic manipulative treatment (OMT) on sacral base asymmetry as assessed by ultrasound. The study will be conducted between July 2016 - June 2017 with data collection planned for August and September 2016. Forty men and women ages 20 to 55 years with at least one or more episodes of LBP in the past two weeks will be recruited from the Kirksville area. Participants will be randomly assigned into two groups, control or OMT using a random number generator. Males and females will be randomized separately to ensure equal distribution into the two study groups. Demographics including sex, age, and body mass index (BMI) will be collected on all participants. All participants will complete a brief medical history questionnaire, receive an initial palpatory assessment of the sacral base asymmetry, and then an initial ultrasound evaluation of sacral base asymmetry. After the ultrasound assessment, the control group will wait in another room for approximately 30 minutes. Participants in the OMT group will receive OMT to address sacral base asymmetry after the initial ultrasound assessment. Following the treatment period for the OMT group, all participants will receive a second ultrasound assessment of sacral base asymmetry. The ultrasonographer will be blinded on whether the subject received an OMT or not. After the second ultrasound measurement, the participants in the control group will be offered an OMT treatment consistent with that of the OMT group.

ELIGIBILITY:
Inclusion Criteria:

Must have experienced at least one or more episodes of LBP in the past two weeks Must be able to lie prone for 30 minutes Must be able to tolerate OMT -

Exclusion Criteria:

Prior spinal surgery Fractures Known congenital anomalies of the lumbar vertebra and sacrum Cannot lie prone for 30 minutes Cannot tolerate OMT

-

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Change in Sacral Base Asymmetry with OMT | Immediately pre and post treatment - approximately 30 minutes between measurements
  Determine the extent to which OMT affects the relative asymmetry between the pelvic and sacral landmarks as measured by ultrasonography when compared to control group.

SECONDARY OUTCOMES:
Change in Sacral Base Asymmetry without OMT | 30 minutes between measurements
  Determine if ultrasound measurements of sacral landmarks are stable over 30 minutes in untreated (control) participants.

OTHER OUTCOMES:
Agreement between palpatory and ultrasound measurements | Approximately 10 mins between palpatory and ultrasound measurements
  Determine if ultrasound measurements of sacral base asymmetry agree with palpatory assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Karen T Snider, DO, FAAO, Principal Investigator — A.T. Still University
Locations (1):
- A.T. Still University, Kirksville, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lockwood MD, Kondrashova T, Johnson JC. Feasibility of Using Ultrasonography to Establish Relationships Among Sacral Base Position, Sacral Sulcus Depth, Body Mass Index, and Sex. J Am Osteopath Assoc. 2015 Nov;115(11):648-53. doi: 10.7556/jaoa.2015.135. PMID 26501757
- [Derived] Snider KT, Redman CL, Edwards CR, Bhatia S, Kondrashova T. Ultrasonographic Evaluation of the Effect of Osteopathic Manipulative Treatment on Sacral Base Asymmetry. J Am Osteopath Assoc. 2018 Mar 1;118(3):159-169. doi: 10.7556/jaoa.2018.035. PMID 29480916

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-01-08): https://cdn.clinicaltrials.gov/large-docs/01/NCT02820701/Prot_SAP_000.pdf
  • Informed Consent Form (2019-01-08): https://cdn.clinicaltrials.gov/large-docs/01/NCT02820701/ICF_001.pdf